CLINICAL TRIAL: NCT02661659
Title: A Phase Ib Trial of a Maintenance Multipeptide Vaccine (S-588210) in Patients With Unresectable Malignant Pleural Mesothelioma Without Progression After First-Line Chemotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI stopped study due to inability to accrue.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-1519
Record Dates: First submitted 2016-01-20; First posted 2016-01-22 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Malignant Pleural Mesothelioma (MPM)
Keywords: mesothelioma; multipeptide vaccine; S-588210
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly Vaccination (Other): Maintenance multipeptide vaccine (S-588210) administered every week
  Interventions: Biological: Multipeptide vaccine S-588210
- Every other Week Vaccination (Other): Maintenance multipeptide vaccine (S-588210) administered every other week
  Interventions: Biological: Multipeptide vaccine S-588210

INTERVENTIONS:
Biological: Multipeptide vaccine S-588210

SUMMARY:
A phase Ib study investigating the safety, the immunogenicity and the optimal administration frequency of the S-588210 5-peptide vaccine in MPM patients without progression after pemetrexed-based chemotherapy will be conducted. Additionally, to identify more accurate predictive biomarkers of response to S-588210, T-cell-receptor-sequencing (TCR) pre- and post-vaccination will be performed in blood samples of patients treated with the vaccine. Immunohistochemical analysis of the vaccine oncoantigens will also be correlated with induction of antigen-specific T-cell responses. Finally, to explore the infiltration of tumors with T-cells and the potential presence of an immunosuppressive tumor microenvironment, immunohistochemistry for immune checkpoints (including PDL1/PD1, CTLA4) and immune suppressive cell subsets (T-regs, macrophages) will be performed.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the rate of peptide-specific CTL induction to S-588210 within the first 8 months in HLA-A*02:01-positive patients with MPM who have not progressed on first-line pemetrexed-based chemotherapy treated on a weekly or every other week vaccination schedule.

Secondary Objectives:

1. To evaluate the safety of S-588210 in HLA-A*02:01-positive patients with MPM treated with S-588210
2. To determine the disease control rate (DCR) in HLA-A*02:01-positive patients with MPM treated with S-588210
3. To determine the progression-free-survival (PFS) in HLA-A*02:01-positive patients with MPM who have not progressed on first-line pemetrexed-based chemotherapy and who are treated with S-588210
4. To evaluate the peptide-specific CTL response to S-588210 over time up to 8 months in HLA-A*02:01-positive patients with MPM who have not progressed on first-line pemetrexed-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable MPM that have completed 4-6 cycles of standard first-line pemetrexed-based chemotherapy for at least 1 month and have not progressed
* Age>18
* Able to provide informed consent for the study
* HLA-A*02:01 positive
* ECOG PS=0-1 at enrollment
* Measurable indicator lesion by modified RECIST criteria
* Adequate bone marrow (ANC > 1000cells/ml, PLT > 50,000/ml, Hg > 8gr/dL), renal (Cr > 2.5xUNL) and liver function (AST, ALT< 3x UNL, total bilirubin < 2x UNL, ALP < 3x UNL)
* Archival tumor tissue available for IHC (1 paraffin-embedded block)
* Epithelioid or biphasic histology

Exclusion Criteria:

* Chemotherapy or investigational antineoplastic drug within 1 month of planned initiation of vaccine therapy
* Patients who received DEPDC1, MPHOSPH1, URLC10, CDCA1, or KOC1 peptide vaccines before
* Active treatment with corticosteroids or other immunosuppressive agents
* Patients who are expected to require any of the following therapies between enrollment and completion or discontinuation of the study treatment:

  1. immunosuppressive drugs, including corticosteroids, methotrexate, mercaptopurine, azathioprine, cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, ATG (anti-thymoglobulin), IL2-receptor antibodies (basiliximab, daclizumab), TNF-a antibodies (infliximab, etanercept, adalimumab)
  2. radiotherapy for the target disease
  3. surgical therapy for the target disease
* History of bone marrow transplantation
* Active infection
* Human immunodeficiency virus infection
* History of or active systemic autoimmune disorder or immunodeficiency syndromes
* History of severe (CTCAE v.4.03 grade 3 or higher) allergic reaction to a drug, vaccination, or biological preparation.
* Pregnancy
* Patients who cannot or do not intend to practice effective contraception
* Severe illness requiring hospitalization
* Lymphocytes <15% of total WBCs at baseline
* Sarcomatoid histology
* Severe (CTCAE v.4.03 grade 3 or higher) concurrent hepatic impairment, renal impairment, heart disease, hematological disease, respiratory disease, or metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who show in vitro cytotoxic T lymphocyte induction to at least 2 of the 5 antigens determined by Enzyme-Linked ImmunoSpot (ELISPOT) assay | Within 8 months from initiation of vaccination

SECONDARY OUTCOMES:
Toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v4.03 | Up to 4 weeks
Disease control rate defined as the proportion of patients who are assessed as having complete response (CR), partial response (PR), or stable disease (SD) (>3 months) | 6 months
6-month progression-free survival (PFS) rate | 6 months
Peptide-specific cytotoxic T lymphocyte response determined by Enzyme-Linked ImmunoSpot (ELISPOT) assay | At 2, 3, 4, 6 and 8 months of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States